CLINICAL TRIAL: NCT02773732
Title: A Phase Ib/II Clinical Trial of Oral Ciprofloxacin and Etoposide in Subjects With Resistant Acute Myeloid Leukemia (AML)
Brief Title: Clinical Trial of Oral Ciprofloxacin and Etoposide in Subjects With Resistant Acute Myeloid Leukemia (AML)(UF-AML-CE-101)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600693; UF-AML-CE-101 (Other: University of Florida); OCR14651 (Other: OF OnCore)
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Leukemia; Acute Myelogenous Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Ciprofloxacin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ciprofloxacin Dose Level 0 (Experimental)
  Interventions: Drug: Ciprofloxacin 750 MG; Drug: Etoposide
- Ciprofloxacin Dose Level +1 (Experimental)
  Interventions: Drug: Etoposide; Drug: Ciprofloxacin 1000 MG
- Ciprofloxacin Dose Level -1 (Experimental)
  Interventions: Drug: Etoposide; Drug: Ciprofloxacin 500 mg

INTERVENTIONS:
Drug: Ciprofloxacin 750 MG — 750 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Other Names: Cipro
  Arms: Ciprofloxacin Dose Level 0
Drug: Etoposide — Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
  Other Names: VP-16; Vepesid
Drug: Ciprofloxacin 1000 MG — 1000 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Other Names: Cipro
  Arms: Ciprofloxacin Dose Level +1
Drug: Ciprofloxacin 500 mg — 500 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Other Names: Cipro
  Arms: Ciprofloxacin Dose Level -1

SUMMARY:
The purpose of the first part of this study is to establish the maximum tolerated dose (MTD) of oral ciprofloxacin when given in combination with a fixed dose of oral etoposide in patients with resistant acute myeloid leukemia (AML). The purpose of the second part of this study is to determine if the established dose of oral ciprofloxacin in combination with oral etoposide is effective in the treatment of patients with resistant AML.

DETAILED DESCRIPTION:
This study will look at: any side effects that occur, the effectiveness of the study drug, and how your disease reacts to ciprofloxacin in combination with etoposide. This study will try to find the highest tolerated dose of ciprofloxacin without causing serious side effects.

Ciprofloxacin is a commonly used antibiotic drug that is approved for use by the United States Food and Drug Administration (FDA). The FDA has not approved ciprofloxacin to treat AML. Etoposide is an anticancer chemotherapy drug that is approved for use by the FDA for the treatment of small cell lung cancer and testicular cancer. Etoposide is also used for treatment of various blood cancers.

There is laboratory research that has shown that ciprofloxacin can make leukemia cells more sensitive to etoposide chemotherapy. This observation indicates that ciprofloxacin may help improve the effectiveness of etoposide in the treatment of resistant AML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML confirmed by review of bone marrow pathology at the University of Florida.
* Patients with relapsed and /or refractory AML who: failed to achieve complete remission (CR) or complete remission with incomplete blood count recovery (CRi) after at least one cycle of induction chemotherapy and not suitable for a second cycle of standard intensive chemotherapy; or who have progressed after 1 cycle of hypomethylating agent or intolerant to hypomethylating agent therapy and not suitable for standard induction chemotherapy regimens; or have relapsed after any duration of response.
* Per the treating physician, the subject must have a life expectancy of >= 4 weeks.
* Subject performance status must be Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2.
* Subject must have a total bilirubin <= 2 mg/dL and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 times the upper limit of normal.
* Subject must have serum creatinine < 2 mg/dL.
* Females of child-bearing potential may participate, provided they meet the following conditions: Must agree to use physician-approved contraceptive methods throughout the study and for 6 months following the last dose of ciprofloxacin and/or etoposide; Must have a negative serum pregnancy test within 7 days prior to beginning treatment on this study.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods throughout the study and should avoid conceiving children for 6 months following the last dose of ciprofloxacin and/or etoposide.
* Must provide written informed consent and be willing to comply with all study-related procedures.

Exclusion Criteria:

* History of allergic or significant adverse reaction [e.g., anaphylaxis, prolonged QTc, or severe tendonitis] to ciprofloxacin or etoposide.
* Acute promyelocytic leukemia (APL) with t(15;17).
* Prolonged baseline QTc, defined as QTc interval > 470 msec in women and > 450 msec in men, or > 480 msec in subjects with a bundle branch block.
* Uncontrolled, clinically significant infection. Subjects with a fever (temperature >= 38.3) thought to be related to leukemia are eligible assuming that blood cultures are negative during the 7 days prior to Cycle 1 Day 1 and there is no clinical evidence of active infection (e.g., negative or stable radiographs and negative physical examination).
* Ongoing, symptomatic Clostridium difficile infection. Subjects who are asymptomatic with negative stool for C. difficile may participate.
* Pregnant and or nursing.
* History of Myasthenia Gravis.
* Treatment with any anticancer therapy (standard or investigational) within 14 days prior to the first dose of ciprofloxacin or less than full recovery from the clinically significant toxic effects of that treatment. The use of hydroxyurea is allowed only during the first 14 days of Cycle 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Brown, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Cancer Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gera K, Cline C, Al-Mansour Z, Medvec A, Lee JH, Galochkina Z, Hsu J, Hiemenz J, Farhadfar N, Dean EA, Wingard JR, Brown R. A phase ib clinical trial of oral ciprofloxacin and etoposide in subjects with resistant acute myeloid leukemia. Leuk Lymphoma. 2024 Oct;65(10):1502-1510. doi: 10.1080/10428194.2024.2361111. Epub 2024 Jun 6. PMID 38841781

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin Dose Level 0: 750 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
- Ciprofloxacin Dose Level +1: 1000 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
Period: Ciprofloxacin Dose Level 0
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Ciprofloxacin Dose Level +1
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
Started | 0 | 8
Completed | 0 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1 | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 68.67 [61 to 75] | 61.75 [21 to 80] | 63.64 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 5 | 7
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Establish the maximum tolerated dose (MTD) of oral ciprofloxacin when given in combination with a fixed dose of oral Etoposide for the treatment of resistant AML.
Time Frame: 1 month
Population: 2 subjects were not evaluable for this outcome measure.
Measure: Number; unit: milligrams
Groups:
- Ciprofloxacin and Etoposide: Ciprofloxacin: Ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Dose Level 0 Ciprofloxacin 750 mg Dose Level +1 Ciprofloxacin 1000 mg Dose Level -1 Ciprofloxacin 500 mg
  Etoposide: Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
Arm/Group | Ciprofloxacin and Etoposide
Number analyzed (Participants) | 9
milligrams | 1000

2. Primary Outcome: Rate of Complete Remission
Description: Determine the rate of complete remission (CR) following treatment with the MTD of oral ciprofloxacin in combination with oral Etoposide for the treatment of resistant AML.
Time Frame: 0 months
Population: No participants were analyzed for this outcome measure because the study did not proceed to phase II.
Arm/Group | Ciprofloxacin and Etoposide
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Duration
Description: Measure the response duration following treatment with oral ciprofloxacin in combination with oral etoposide for the treatment of resistant AML.
Time Frame: 111 days
Population: Only 1 participant in the ciprofloxacin Dose Level +1 cohort had a response to measure response duration.
Measure: Number; unit: days
Arm/Group | Ciprofloxacin Dose Level +1
Number analyzed (Participants) | 1
days | 111

4. Secondary Outcome: Progression-free Survival
Description: Measure progression-free survival following treatment with oral ciprofloxacin in combination with oral Etoposide for the treatment of resistant AML.
Time Frame: 317 days
Measure: Mean (Full Range); unit: days
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
Number analyzed (Participants) | 3 | 8
days | 56 [25 to 115] | 92.25 [26 to 317]

5. Secondary Outcome: Overall Survival
Description: Measure overall survival following treatment with oral ciprofloxacin in combination with oral Etoposide for the treatment of resistant AML.
Time Frame: 317 days
Population: 1 subject was still alive at the time protocol follow-up was discontinued, so they are not included in the analysis for this outcome measure.
Measure: Mean (Full Range); unit: days
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
Number analyzed (Participants) | 3 | 7
days | 140.67 [25 to 282] | 109.29 [43 to 317]

6. Secondary Outcome: Percentage of Grade ≥ 3 Adverse Events
Description: Estimate the rate of Grade ≥ 3 adverse events following treatment with oral ciprofloxacin and oral etoposide at the MTD.
Time Frame: 93 days
Measure: Number; unit: percentage of reported adverse events
Groups:
- Ciprofloxacin Dose Level 0: 750 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Etoposide: Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
- Ciprofloxacin Dose Level +1: 1000 mg ciprofloxacin will be taken orally twice daily on Days 1 to 10 of each 28-day cycle.
  Etoposide: Etoposide 200 mg will be taken orally once daily on Days 2 to 8 of each 28-day cycle.
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
Number analyzed (Participants) | 3 | 8
percentage of reported adverse events | 20 | 28.45

ADVERSE EVENTS:
Time Frame: At minimum, adverse event data were collected at screening, every 7 days during study treatment and at 28 days after the last dose of study treatment. Adverse event data were collected for a maximum of 93 days for all participants. All-cause mortality data was collected over a maximum of 317 days for all participants.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator at screening, every 7 days during study treatment, and at 28 days after the last dose of study treatment at a minimum. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Ciprofloxacin Dose Level 0 | Ciprofloxacin Dose Level +1
All-Cause Mortality (participants affected / at risk) | 3/3 | 7/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin Dose Level 0 (N=3) | Ciprofloxacin Dose Level +1 (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Cardiac disorders - other, specify (Cardiac disorders) | 1 | 0 — cardiogenic shock
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Metabolism and nutrition disorders - other, specify (Metabolism and nutrition disorders) | 0 | 1 — failure to thrive
Encephalopathy (Nervous system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin Dose Level 0 (N=3) | Ciprofloxacin Dose Level +1 (N=8)
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Cardiac disorders - other, specify (Cardiac disorders) | 0 | 1 — systolic murmur
Chills (General disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Eye pain (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 2 | 4
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 0 | 1 — indigestion
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 0 | 1 — loose stool
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 0 | 1 — C. diff infection
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 5
Hypotension (Vascular disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 1 — hyperphosphatemia
Investigations - Other, specify (Investigations) | 0 | 1 — total protein decreased
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 3
Mucosal infection (Infections and infestations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 — musculoskeletal pain bilateral legs and arms
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 — acute renal insufficiency
Sinus tachycardia (Cardiac disorders) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 — perirectal irritation
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
White blood cell decreased (Investigations) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT02773732/Prot_SAP_000.pdf